CLINICAL TRIAL: NCT03773822
Title: Low Dose of Hydrocortisone and Fludrocortisone in Adult Cardiogenic Shock. A Multicenter, Prospective, Double-blind, Randomized, Placebo-controlled Study
Brief Title: Low Dose of Hydrocortisone and Fludrocortisone in Adult Cardiogenic Shock.
Acronym: COCCA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018/05
Record Dates: First submitted 2018-11-21; First posted 2018-12-12 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Cardiogenic Shock
Keywords: Cardiogenic Shock; Steroids; Hydrocortisone; Fludrocortisone; Reversal of shock; Mortality; Adrenal insufficiency
MeSH Terms: conditions — Shock, Cardiogenic; Adrenal Insufficiency | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo of hydrocortisone and placebo of fludrocortisone (Placebo Comparator): Placebo of hydrocortisone as an iv bolus every 6 hours for seven days plus placebo of enteral fludrocortisone given once a day for seven days
  Interventions: Other: Placebo
- Combination of hydrocortisone + fludrocortisone (Experimental): Hydrocortisone will be given as 50 mg iv bolus every 6 hours for seven days and a tablet of 50 µg of fludrocortisone will be given once a day enterally for seven days
  Interventions: Combination Product: Hydrocortisone + Flucortac

INTERVENTIONS:
Combination Product: Hydrocortisone + Flucortac — Low dose steroids
  Arms: Combination of hydrocortisone + fludrocortisone
Other: Placebo — Placebo
  Arms: Placebo of hydrocortisone and placebo of fludrocortisone

SUMMARY:
The purpose of this randomized controlled trial is to evaluate the hemodynamic effect of low dose corticosteroid therapy (hydrocortisone and fludrocortisone) in the treatment of adult cardiogenic shock.

DETAILED DESCRIPTION:
Cardiogenic shock is a serious condition with a high mortality rate, characterized by acute dysfunction of the heart pump. Critical illness-related corticosteroid insufficiency is a pathophysiological concept, first described in septic shock. It is characterized by an impairment of the hypothalamic pituitary axis during critical illness. Its diagnosis is usually suggested by an inappropriate response to the adrenal stimulation test. The results of corticosteroid supplementation studies in septic shock are controversial, but most of these studies demonstrate that corticosteroid therapy improves reversal of shock.

The concept of critical illness-related corticosteroid insufficiency has recently been expanded to cardiogenic shock. The latter has many physiopathological similarities with septic shock. However, no studies have evaluated the effect of supplemental corticosteroid supplementation in cardiogenic shock.

The purpose of this study is to evaluate the hemodynamic effect of low dose corticosteroid therapy in the treatment of adult cardiogenic shock.

This study is a multicenter, randomized, double blinded, placebo controlled trial comparing intravenous hydrocortisone (50 mg intravenously every 6 hours) plus enteral fludrocortisone (50 µg/day) with placebo for seven days in critically ill patients with cardiogenic shock.

The primary endpoint for this trial will be catecholamine-fee days at day-7. Secondary endpoints will include all-cause mortality at 28 and 90 days after randomisation.

Several pre-defined sub-groups analyses are planned, including: postcardiotomy, myocardial infarction, etomidate use, vasopressor use...

380 patients will be enrolled in this study at approximately 20 study sites. Each patient will be followed-up for 90 days.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years
2. Cardiogenic shock state, according to the consensual definition:

   1. Systemic arterial hypertension (systolic blood pressure <90 mmHg or mean arterial pressure ≤ 65 mmHg) or signs of peripheral hypoperfusion, requiring treatment with catecholamines to maintain systolic blood pressure ≥ 90 mmHg and regression of signs of hypoperfusion;
   2. Presence of at least one sign of systemic hypoperfusion among the following: marbling, oliguria ≤ 25 ml / h, impairment of consciousness, arterial hyperlactatemia> 2 mmol / L;
   3. Presence of at least one sign of hypocontractility or low flow among the following: cardiac index ≤ 2.2 L / min / m2, left ventricular ejection fraction (LVEF) ≤ 40% or full time velocity (ITV) under aortic ≤ 18 cm, or need for catecholamines to maintain an index
   4. Clinical signs of left and / or right cardiac congestion (clinical sign of acute cardiogenic pulmonary edema or jugular turgor or edema of the lower limbs), radiological (bilateral alveolar opacities compatible with acute cardiogenic pulmonary edema), echocardiography (elevation of filling pressures of the left ventricle measured with Doppler: E / A> 2 if LVEF ≤40% or E / Ea> 13 if LVEF> 40%; or estimated PAPS> 35mmHg) or with right cardiac catheterization (pulmonary artery occlusion pressures> 15mmHg or PAPm> 25mmHg)
3. Having received informed information about the study and having signed a consent to participate in the study
4. Benefiting from a social security

Exclusion Criteria:

1. Cardiogenic shock state with catecholamine infusion for more than 24 hours;
2. Presence Presence of septic shock at inclusion;
3. Cardiopulmonary arrest recovered in the 7 days preceding inclusion with at least one early sign of poor prognosis among the following: no control, non-shockable rhythm, CAHP score (Cardiac Arrest Hospital Prognosis)> 150;
4. Patients already on circulatory support (ECMO) before inclusion (patients who are assisted after inclusion will not be excluded);
5. Cardiogenic shock on viral myocarditis;
6. Prior corticosteroid therapy (≥ 30 mg prednisone or equivalent ≥ 1 month);
7. Receiving one of the following treatments: ketoconazole, rifampicin, phenytoin, phenobarbital, cyclosporine and clarithromycin;
8. Known history of hypersensitivity to fludrocortisone or hydrocortisone;
9. Known pregnancy or breastfeeding;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Patients not treated with corticosteroids at day 7 | 7 days

SECONDARY OUTCOMES:
Mortality at 28 and 90 days after randomisation | 28 and 90 days after randomisation
Modification of the cardiac index | 7 days
Length of stay in intensive care and hospital | 28 and 90 days after randomisation
Duration of support by catecholamines | 28 days after randomisation
Clearance of lactatemia | 7 days
Number of patients use of mechanical ventilation | 28 days after randomisation
Number of patients with Circulatory assistance | 28 days after randomisation
Number of patients alive at day 7 without failure (SOFA) score) | 7 days
Rate of patients with nosocomial infection | 28 days after randomisation
Rates of patients requiring the introduction of intravenous insulin therapy after randomization | 7 days
Modification of mean arterial pressure | 7 days

CONTACTS AND LOCATIONS:
Locations (21):
- France (21):
  - Hôpital Parly II, Le Chesnay, Le Chasnay
  - CH Intercommunal de Villeneuve Saint Georges, Villeneuve-Saint-Georges, Villeneuve Saint Georges
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - CH de Marne la Vallée - Site Jossigny, Jossigny
  - CHU Lille - Institut Cœur Poumon, Lille
  - Centre Hospitalier Saint Joseph Saint Luc, Lyon
  - Hôpital Privé Jacques Cartier, Massy
  - Hôpital Arnaud-de-Villeneuve, Montpellier
  - CMC Ambroise Paré, Neuilly-sur-Seine
  - CHU de Nîmes, Nîmes
  - Hôpitaux Universitaires Pitié Salpêtrière, Paris
  - Groupe Hospitalier Paris Saint Joseph, Paris
  - Hôpital Cochin, Paris
  - Hôpital européen Georges-Pompidou, Paris
  - Hôpital Bichat, Paris
  - CH Pontoise, Pontoise
  - Centre cardiologique du nord saint denis, Saint-Denis
  - CHU de Strasbourg, Strasbourg
  - Hopital Rangueil, Toulouse
  - CHRU Hôpitaux de Tours, Tours
  - Hôpital Henri Mondor, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mekontso Dessap A, Bagate F, Delmas C, Morichau-Beauchant T, Cholley B, Cariou A, Lattuca B, Moussa M, Mongardon N, Fard D, Schmidt M, Bougle A, Kerneis M, Vivier E, Roubille F, Duprey M, Decalf V, Genet T, Merzoug M, Audureau E, Squara P. Low-dose corticosteroid therapy for cardiogenic shock in adults (COCCA): study protocol for a randomized controlled trial. Trials. 2022 Jan 3;23(1):4. doi: 10.1186/s13063-021-05947-6. PMID 34980224